CLINICAL TRIAL: NCT01697644
Title: Growth Hormone Treatment of Children After Intrauterine Growth Retardation
Brief Title: Growth Hormone Treatment of Children Diagnosed of Intrauterine Growth Retardation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHRETARD/NL/21
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Experimental)
  Interventions: Drug: somatropin
- High dose (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 3 IU/m^2/day. Dose adjusted approximately every 3 months. Injected subcutaneously once daily
  Arms: Low dose
Drug: somatropin — 3 IU/m^2/day. Dose adjusted approximately every 3 months. Injected subcutaneously once daily
  Arms: High dose

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess and compare the efficacy and safety of two dose levels of somatropin over a long period (till final height is reached). This trial is an extension to trials GHRETARD/BDP/14/NL (a 2-year initial trial) and GHRETARD/BPD/20/NL (a 2-year extension trial).

ELIGIBILITY:
Inclusion Criteria:

* Completion of the GHRETARD/BPD/20/NL trial
* Written informed consent from child and/or parents/guardians before continuation in the extension trial

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 1990-10; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Linear growth (height during childhood)
Final height
Bone maturation
Pubertal development

SECONDARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry B. (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Rotterdam, Netherlands

REFERENCES:
- [Result] Boonstra V, van Pareren Y, Mulder P, Hokken-Koelega A. Puberty in growth hormone-treated children born small for gestational age (SGA). J Clin Endocrinol Metab. 2003 Dec;88(12):5753-8. doi: 10.1210/jc.2003-030512. PMID 14671164
- [Result] Sas T, de Waal W, Mulder P, Houdijk M, Jansen M, Reeser M, Hokken-Koelega A. Growth hormone treatment in children with short stature born small for gestational age: 5-year results of a randomized, double-blind, dose-response trial. J Clin Endocrinol Metab. 1999 Sep;84(9):3064-70. doi: 10.1210/jcem.84.9.5942. PMID 10487666
- [Result] Sas T, Mulder P, Hokken-Koelega A. Body composition, blood pressure, and lipid metabolism before and during long-term growth hormone (GH) treatment in children with short stature born small for gestational age either with or without GH deficiency. J Clin Endocrinol Metab. 2000 Oct;85(10):3786-92. doi: 10.1210/jcem.85.10.6917. PMID 11061539
- [Result] Sas TC, Gerver WJ, De Bruin R, Mulder PG, Cole TJ, De Waal W, Hokken-Koelega AC. Body proportions during 6 years of GH treatment in children with short stature born small for gestational age participating in a randomised, double-blind, dose-response trial. Clin Endocrinol (Oxf). 2000 Dec;53(6):675-81. doi: 10.1046/j.1365-2265.2000.01155.x. PMID 11155088
- [Result] Sas T, Mulder P, Aanstoot HJ, Houdijk M, Jansen M, Reeser M, Hokken-Koelega A. Carbohydrate metabolism during long-term growth hormone treatment in children with short stature born small for gestational age. Clin Endocrinol (Oxf). 2001 Feb;54(2):243-51. doi: 10.1046/j.1365-2265.2001.01178.x. PMID 11207640
- [Result] Van Pareren Y, Mulder P, Houdijk M, Jansen M, Reeser M, Hokken-Koelega A. Adult height after long-term, continuous growth hormone (GH) treatment in short children born small for gestational age: results of a randomized, double-blind, dose-response GH trial. J Clin Endocrinol Metab. 2003 Aug;88(8):3584-90. doi: 10.1210/jc.2002-021172. PMID 12915640
- [Result] van Pareren Y, Mulder P, Houdijk M, Jansen M, Reeser M, Hokken-Koelega A. Effect of discontinuation of growth hormone treatment on risk factors for cardiovascular disease in adolescents born small for gestational age. J Clin Endocrinol Metab. 2003 Jan;88(1):347-53. doi: 10.1210/jc.2002-020458. PMID 12519875
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com